CLINICAL TRIAL: NCT03830710
Title: Detection of Salivary 8-Hydroxy-2-Deoxyguanosine and Total Antioxidant Capacity in Patients With Oral Premalignant and Malignant Lesions
Brief Title: 8-Hydroxy-2-Deoxyguanosine ,Total Antioxidant Capacity in Oral Premalignant and Malignant Lesions
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Sandy Hassan, lecturer, Fayoum University
Other Study IDs: 1234
Record Dates: First submitted 2019-01-28; First posted 2019-02-05 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Premalignant Lesion
Keywords: Squamous cell carcinoma; 8-hydroxy-2- deoxyguanosine; Antioxidant
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group A: 30 patients diagnosed with oral leukoplakia
- Group B: 30 patients diagnosed with oral lichen planus
- Group C: 30 patients having oral squamous cell carcinoma with the tongue being the most commonly affected site
- Group D: 30 age and gender matched individuals having no oral mucosal lesions acting as a control group

SUMMARY:
Objectives: Investigating the level of salivary 8-hydroxy-2-deoxyguanosine (8-OHdG) and total antioxidant capacity (TAC) in oral premalignant and malignant lesions in order to determine their diagnostic value for the malignant patients. Design: 120 subjects diagnosed with oral leukoplakia, oral lichen planus (OLP) and oral squamous cell carcinoma (OSCC) along with healthy control subjects were included. Salivary samples from all participants were collected. 8-OHdG was measured by ELISA technique and the TAC level was assessed by a photometric test system.

DETAILED DESCRIPTION:
Detection of molecular markers in saliva is superior to their detection in serum and other body fluids due to the fact of being an easy non-invasive tool requiring no training for its collection. Consequently, the aim of our work was to investigate salivary 8-OHdG and TAC in premalignant and malignant patients compared to normal subjects and to determine their diagnostic value for the malignant patients.

Methodology:

Study population:

A total of 120 subjects were enrolled in the present study. The clinically tested and confirmed subjects included Group A: 30 patients diagnosed with oral leukoplakia Group B: 30 patients suffering from oral lichen planus Group C: 30 patients having oral squamous cell carcinoma with the tongue being the most commonly affected site Group D: 30 age and gender matched individuals having no oral mucosal lesions acting as a control group.

Comprehensive oral diagnosis was done for all participating individuals. Biopsy specimens were obtained from various lesions where a surgical double wedge incisional biopsy was carried out to a depth of about 2mm. Specimens were sent for histopathological examination to confirm the clinical diagnosis.

Salivary sample collection: Collection of whole unstimulated saliva from all participants was performed using standard techniques.Subjects refrained from eating, drinking, chewing gum etc., for at least ½ h before the evaluation.Samples were collected by asking individuals to swallow first, tilt their head forward and expectorate all saliva in a tube for 5 minutes without swallowing. After collection, all samples were immediately stored at -20ºC until assayed.

Detection of salivary 8-OHdG: Saliva was centrifuged for 5 minutes at 5000 x g. The supernatant was removed for determination of 8- hydroxy-2'-deoxyguanosine using an ELISA kit provided by BioVision, USA (Catalog # K4160-100). 8-hydroxy-2'-deoxyguanosine is an oxidized derivative of deoxyguanosine and is one of the major products of DNA oxidation.

Determination of salivary total antioxidative status/capacity (TAS/TAC) was done using ImAnOx (TAS/TAC) Kit provided by Immun Diagnostik, Germany. It is a photometric test system used for the determination of the total antioxidative status/capacity in EDTA-plasma, serum and other biological samples.

The determination of the antioxidative capacity was performed by the reaction of antioxidants in the sample with a defined amount of exogenously provided hydrogen peroxide (H2O2). The antioxidants in the sample eliminate a certain amount of the provided H2O2. The residual H2O2 was determined photometrically by an enzymatic reaction which involves the conversion of TMB to a colored product. After addition of a stop solution, the samples were measured at 450 nm in a microtiter plate reader. The quantification was performed by the delivered calibrator. The difference between applied and measured peroxide concentration in a defined time period is proportional to the reactivity of the antioxidants of the sample (antioxidative capacity). Quantification was performed with the enclosed calibrator.

ELIGIBILITY:
Inclusion Criteria:

All included individuals were not under any current medication, suffering from any systemic condition or having any other oral mucosal disorder.

Exclusion Criteria:

1. Pregnant or lactating females
2. subjects having systemic disorder or taking medications;
3. subjects who suffer from any other mucosal lesions.
4. severe periodontal inflammation

Ages: 35 Years to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The included subjects were all assessed medically according to the modified Cornell Medical index (Kerr & Millard, 1965).
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Salivary 8-OHdG | 1 year
  8-OHdG have a critical role in the pathogenesis of malignant lesions
salivary TAC | 1 year
  OSCC might be used as a tool to help diagnosis of OSCC but not to differentiate between various malignant grades

CONTACTS AND LOCATIONS:
Locations (1):
- Sandy hassan shaaban, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-04-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT03830710/SAP_000.pdf